CLINICAL TRIAL: NCT03931655
Title: A Preliminary Study of Photoacoustic Imaging to Detect Micrometastases in the Lymph Nodes of Breast Cancer Patients
Brief Title: Photoacoustic Lymph Node Imaging
Status: Terminated | Type: Observational
Why Stopped: There have been multiple issues getting the device repaired and then in working order. The PI's have decided to terminate the study. The termination request has been filed with the institution's IRB.
Sponsor: Geoff Luke (Other)
Collaborators: Dartmouth College (Other); Dartmouth-Hitchcock Medical Center (Other)
Responsible Party: Sponsor-Investigator, Geoff Luke, Co-Investigator and Regulatory Sponsor, Dartmouth-Hitchcock Medical Center
Organization: Dartmouth-Hitchcock Medical Center (Other)
Other Study IDs: STUDY00031569; D18155 (Other: Dartmouth College)
Record Dates: First submitted 2019-04-15; First posted 2019-04-30 (Actual); Last update posted 2023-11-07 (Actual); Status verified 2023-11

CONDITIONS: Breast Cancer
Keywords: Photoacoustic imaging; Lymph nodes; micrometastases
MeSH Terms: conditions — Breast Neoplasms; Neoplasm Micrometastasis

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Spectroscopic photoacoustic imaging: Any suspicious lymph nodes identified through ultrasound will be imaged with spectroscopic photoacoustic imaging, which is a diagnostic test to measure saturated oxygen in the nodes.
  Interventions: Diagnostic Test: Spectroscopic photoacoustic imaging

INTERVENTIONS:
Diagnostic Test: Spectroscopic photoacoustic imaging — Spectroscopic photoacoustic imaging uses a laser that is pulsed for a nanosecond, applying laser light to the patient's skin. Hemoglobin and melanin absorb the laser's energy and convert it to heat, which rapidly expands local tissue and produces a broadband ultrasound wave and is detected with a clinical ultrasound transducer. Because the signal is proportional to the optical absorption in tissue, high resolution images of the lymph nodes can be acquired from the detected ultrasound waves, and can be used to measure saturated oxygen in the nodes.

SUMMARY:
In this spectroscopic photoacoustic imaging study, the investigators will acquire images (only) to:

1. determine if spectroscopic photoacoustic imaging can acquire high fidelity images in a clinical setting,
2. discover if blood oxygen saturation changes are observable in breast cancer patients during early stages of metastatic invasion, and
3. compare the sensitivity and specificity of photoacoustic imaging with ultrasound imaging for the detection of lymph node metastases.

The results from imaging will not be used in any decision making process. This study is solely used to test the photoacoustic imaging device and evaluate it against the current standard of care. The device is completely noninvasive and uses only safe levels of energy as determined by the American National Standards Institute (ANSI) and the FDA. The device does not pose a serious to the health, safety, or welfare of the patient.

DETAILED DESCRIPTION:
The study is centered on determining whether photoacoustic imaging of blood oxygen saturation can detect lymph node metastases.

Patients who are returning for an ultrasound exam after detection of a suspicious node via magnetic resonance imaging will be enrolled in the study.

Enrolled patients will receive a clinical ultrasound exam, as is the current standard of care. Suspicious nodes will be identified and imaged with combined ultrasound and spectroscopic photoacoustic imaging. Measurements will be acquired with three to five replicates with slightly modified transducer positioning to measure system and intranodal variance of the measurements. One to five contralateral axillary lymph nodes will be imaged to serve as a control and to determine patient-to-patient variability in lymph node saturated oxygen. The distance from the skin to the lymph node will also be measured with ultrasound imaging for each node.

If the ultrasound imaging identifies a suspicious node, patients will undergo ultrasound guided biopsy to confirm the true metastatic state of the nodes. Suspicious nodes will be clipped to facilitate identification at the time of axillary node dissection. During the sentinel node procedure, investigators will use intraoperative photoacoustic imaging to measure the blood oxygenation in the sentinel lymph node immediately prior to its removal. Histology will be performed on all biopsy samples and excised nodes to determine the true metastatic state of the node(s).

ELIGIBILITY:
Inclusion Criteria

1. Subjects are female age 18 or older with breast cancer and who will undergo surgical SLN biopsy/procedure or axillary dissection.
2. Subjects are capable of giving informed consent.

Exclusion Criteria

1. Subjects have had prior surgery in or near the axillary lymph nodes.
2. Subjects are currently undergoing chemotherapy, radiation therapy, hormone therapy, or targeted therapy for the breast cancer.
3. Subjects will be receiving neoadjuvant therapy prior to the surgical sentinel lymph node biopsy.
4. Subjects are homeless persons or have active drug/alcohol dependence or abuse history.
5. Subjects are pregnant or breast-feeding.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Female breast cancer patients who are undergoing axillary surgery to assess lymph node status are eligible to be enrolled.
Sampling Method: Non-Probability Sample
Enrollment: 1 (Actual)
Dates: Start 2019-11-01 (Actual); Primary Completion 2023-11-02 (Actual); Study Completion 2023-11-02 (Actual)

PRIMARY OUTCOMES:
Spectroscopic photoacoustic image acquisition feasibility | Through study completion, an average of 12 weeks
  Determine the feasibility of using spectroscopic photoacoustic imaging to determine the metastatic state of lymph nodes prior to surgery/biopsy by measuring changes in blood oxygen saturation.

SECONDARY OUTCOMES:
Spectroscopic photoacoustic image depth | Day 1, up to 12 weeks after imaging
  Determine the maximum imaging depth that can be reliably achieved with spectroscopic photoacoustic imaging.
Spectroscopic photoacoustic imaging device comparison | Day 1, up to 12 weeks after imaging
  Determine the variance of saturated oxygen measurements acquired with spectroscopic photoacoustic imaging.

CONTACTS AND LOCATIONS:
Overall Officials: Roberta M. diFlorio-Alexander, MD, Principal Investigator — Dartmouth-Hitchcock Medical Center
Locations (1):
- Dartmouth-Hitchcock Medical Center, Lebanon, New Hampshire, United States

IPD SHARING:
Plan to Share IPD: No